CLINICAL TRIAL: NCT04285775
Title: A Novel Device for Surveillance of Vascular Access Sites for Bleeding
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Chionh Chang Yin, Senior Consultant, Changi General Hospital
Other Study IDs: NHIC-I2D-1608124
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Dialysis; Complications; Wound Complication; Catheter Complications; Hemorrhage; Bleeding Wound
Keywords: Dialysis; Catheter; Access; Bleeding; Haemorrhage; Mortality; Monitoring; Detection
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Insertion of Dialysis Catheter: Hospital inpatients planned for dialysis catheter insertion, based on standard clinical care and indications as identified by the primary nephrologist-in-charge.
  Interventions: Device: Application of device which monitors for bleeding - Blood Warning Technology with Continuous Hemoglobin sensor (BWATCH)
- Removal of Dialysis Catheter: Hospital inpatients planned for dialysis catheter removal, based on standard clinical care and indications as identified by the primary nephrologist-in-charge.
  Interventions: Device: Application of device which monitors for bleeding - Blood Warning Technology with Continuous Hemoglobin sensor (BWATCH)

INTERVENTIONS:
Device: Application of device which monitors for bleeding - Blood Warning Technology with Continuous Hemoglobin sensor (BWATCH) — A stand-alone disc-shaped device (approximately 5 cm in diameter and <1 cm thick) which can be placed over dressings. Once switched on and put in place, continuous monitoring for bleeding takes place. Detection occurs in 2 phases. First, the system monitors for the appearance of fluid in the dressing by detecting a change in capacitance. Next, a light sensor differentiates blood from other fluids by detecting that a unique spectrum of light (525nm) is absorbed, a property unique for hemoglobin. The presence of fresh blood triggers a loud alarm, alerting medical staff to attend to the patient. The device can be used over transparent plastic dressings and does not require direct contact with blood.

SUMMARY:
Background Bleeding is often encountered after vascular access procedures for dialysis and fatal episodes of haemorrhage has been reported. A technological solution was sought to monitor for such rare but potentially catastrophic incidents. A novel device, BWATCH, was developed to detect fresh blood from wounds.

Aims The aim of this clinical trial was to evaluate the sensitivity and specificity of the device in detecting bleeding in a clinical environment.

Methods This a prospective, observational study on inpatients who will have a dialysis catheter inserted or removed. The device will be placed over the dressing for at least 6 hours. An alarm will be triggered if the device detects moisture and wavelength of light reflected specific for haemoglobin.

DETAILED DESCRIPTION:
Background

Post-procedural wound hemorrhage is a potential complication following any invasive procedure. In the setting of hemodialysis, with multiple repeated vascular access procedures performed on uremic patients prone to bleeding, post-procedural bleeding would not be infrequent.

Serious adverse events following central venous catheter removal, while rare, were not isolated incidents. The British National Reporting and Learning System, reported 6 incidents of late bleeding following femoral line removal over 3 years. Of these, 3 resulted in deaths and 2 suffered more than one litre of blood loss. The UK Renal Association, British Renal Society and Intensive Care Society subsequently released a recommendation for the safe removal of a temporary femoral dialysis line in 2019. Protocols implemented in some units required an intense period of monitoring every 5-15 minutes in the first 2 hours.

However, frequent monitoring protocols places additional demands on already scarce nursing manpower. As catastrophic bleeding is rare, it is difficult to expect healthcare staff to maintain a consistent high level of vigilance for such a low probability event. The possibility of missed catastrophic bleeding is always present, particularly if the patient is incapacitated and unable to call for assistance.

A technological solution to safely monitor patients for bleeding following catheter removal is needed. Ideally, this technology should also be applicable for other wounds at risk of severe bleeding, for example, after arterial access for coronary angiogram or vascular interventions. There were no commercially available devices which fully met the user requirements, which included ease of use, wireless, compact form factor and specific detection of bleeding with no direct contact with the wound or blood. A compact device was developed

Through a research collaboration between a hospital and a technology and design university, supported by a national innovation grant, a device was developed to monitor wound for bleeding. By the end of 2018, a working prototype - Blood Warning Technology with Continuous Hemoglobin sensor (BWATCH) - was available for first-in-human clinical trials. The technological concept has been presented in electrical engineering conferences. This is a stand-alone disc-shaped device (approximately 5 cm in diameter and <1 cm thick) which can be placed over dressings and continuous monitoring for bleeding will take place. The presence of fresh blood triggers a loud alarm, alerting medical staff to attend to the patient.

Objectives

The primary aim of this clinical trial was to evaluate the sensitivity of the device in detecting bleeding in a clinical environment. The secondary aim is to determine the specificity of the device for actual bleeding (false positive rates).

Materials and Methods

This study has been reviewed and approved by the institutional review board (Singhealth cIRB 2014-2036).

This a prospective, observational study performed in an acute care hospital. Inpatients planned for dialysis catheter insertion or removal based on standard clinical care and indications will be identified fro recruitment.

Consent will be obtained from the patient or their legal representative if cognitively impaired. As part of standard care, the procedurist will secure haemostasis following the procedure and apply a bandage. The investigators will then place the device over the dressing and secure it in place. The device will then be left in-situ for at least 6 hours. Any alarms triggered and bleeding episodes will be documented in a case report form.

For safety, throughout the observation period, routine monitoring and inspection for bleeding by the nurse-in-charge would continue as per hospital clinical protocol.

Baseline demographic data of the patients will be collected. Laboratory test results collected will include the platelet count, international normalized ratio (INR) and partial thromboplastin time (PTT). The use of any anti-coagulation or anti-platelet medication will be recorded.

From the bleeding incidences and device alarm activation rates, the sensitivity and specificity of the device for detection of true bleeding will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Hospital inpatients planned for dialysis catheter insertion or removal, based on standard clinical care and indications as identified by the primary nephrologist-in-charge.

Exclusion Criteria:

* Patients who declined participation, or
* Patients with no legal representatives who were unable to provide consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to an acute care hospital with renal failure requiring dialysis. These patients were planned for dialysis catheter insertion or removal, based on standard clinical care and indications as identified by the primary nephrologist-in-charge.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of bleeding events detected by device | 0 to 6 hours after procedure
  Number of bleeding episodes and detected by the device

SECONDARY OUTCOMES:
Number of False Alarms | 0 till 6 hours after procedure or till alarm triggered (whichever is earlier)
  Number of times the device alarm was triggered with no bleeding is observed.
Number of Missed Bleeding Events | 0 to 6 hours after procedure
  Number of episodes of bleeding but no device alarm was triggered.

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Renal Association, British Renal Society, Intensive Care Society. Patient Safety Alert: response to reported death from blood loss following removal of a temporary femoral dialysis catheter. Nov 29, 2018 [cited Feb 01, 2020]. — https://britishrenal.org/news/response-of-the-renal-association-ra-british-renal-society-brs-and-intensive-care-society-ics-to-a-reported-death-from-blood-loss-following-removal-of-a-temporary-femoral-dialysis-catheter/
- See also: The Renal Association, British Renal Society, Intensive Care Society. Recommendation for the safe removal of a temporary femoral dialysis line. May 31, 2019 [cited Feb 01, 2020]. — https://britishrenal.org/news/recommendation-for-the-safe-removal-of-a-temporary-femoral-dialysis-line/